CLINICAL TRIAL: NCT01232257
Title: Effect of N-acetylcysteine on Hydrogen Sulfide in Chronic Kidney Disease
Brief Title: Effect of N-acetylcysteine (NAC) on Hydrogen Sulfide (H2S) in Chronic Kidney Disease (CKD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: A.C. Abrahams (Other)
Responsible Party: Sponsor-Investigator, A.C. Abrahams, MD, UMC Utrecht
Organization: UMC Utrecht (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H2S-NAC
Record Dates: First submitted 2010-11-01; First posted 2010-11-02 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Kidney Disease; Chronic Kidney Failure; End Stage Kidney Disease; End Stage Renal Disease
Keywords: Chronic kidney disease; Chronic kidney failure; End stage kidney disease; End stage renal disease; Hydrogen sulfide; N-acetylcysteine; Acetylcysteine
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Healthy volunteers (Experimental)
  Interventions: Drug: N-acetylcysteine
- CKD patients (Experimental): Patients with CKD stage 3-4 (GFR 15-60 ml/min)
  Interventions: Drug: N-acetylcysteine
- Hemodialysis patients (Experimental)
  Interventions: Drug: N-acetylcysteine
- Peritoneal dialysis patients (Experimental)
  Interventions: Drug: N-acetylcysteine

INTERVENTIONS:
Drug: N-acetylcysteine — 4 gifts of N-acetylcysteine 600 mg BID

SUMMARY:
Cardiovascular morbidity and mortality is high in CKD patients. Nitric oxide (NO) deficiency plays a crucial role in progression of CKD. This leads to endothelial dysfunction, hypertension, and inflammation. Hydrogen sulfide (H2S) could serve as a backup mechanism for NO deficiency in CKD. N-acetylcysteine (NAC) is a derivate of cysteine and this is the main substrate for H2S production. Therefore, NAC should enable us to stimulate H2S production in humans. Our objective is to investigate the effect of NAC on plasma H2S levels and on markers of oxidative stress, inflammation, and endothelial dysfunction in healthy volunteers, CKD patients, and dialysis patients. We hypothesize that there is an increase in H2S levels after treatment with NAC.

ELIGIBILITY:
Inclusion criteria:

Healthy volunteers:

* Adult (> 18 years and older)
* Healthy, as assessed by medical history, blood pressure, plasma creatinine, and urine dipstick
* No medication use

CKD patient:

* Adult (> 18 years and older)
* CKD stage 3-4 (GFR 15-60 ml/min)

Hemodialysis patient:

* Adult (> 18 years and older)
* Hemodialysis patient

Peritoneal dialysis patient:

* Adult (> 18 years and older)
* Peritoneal dialysis patient

Exclusion criteria:

* Unable to give informed consent
* Hypersensitivity to N-acetylcysteine
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Hydrogen sulfide (H2S) | After 48 hours
  Investigate the effect of N-acetylcysteine on plasma H2S levels and on markers of oxidative stress, inflammation, and endothelial dysfunction in healthy volunteers, CKD patients, and dialysis patients

CONTACTS AND LOCATIONS:
Overall Officials: M C Verhaar, MD, PhD, Principal Investigator — UMC Utrecht; A C Abrahams, MD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Netherlands